CLINICAL TRIAL: NCT04894357
Title: Phenotypic and Site Directed Mutagenesis Analysis on the Impact of V106I in HIV-1 Reverse Transcriptase on Resistance to Doravirine
Brief Title: Impact of V106I on Resistance to Doravirine
Acronym: V106IFC
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental (Other)
Responsible Party: Principal Investigator, Federico García, PhD, Head of Clinical Microbiology, Fundación Pública Andaluza para la Investigación Biomédica Andalucía Oriental
Other Study IDs: HUCSC-V106I
Record Dates: First submitted 2021-05-09; First posted 2021-05-20 (Actual); Last update posted 2021-08-18 (Actual); Status verified 2021-08

CONDITIONS: HIV-1-infection
Keywords: doravirine; resistance; V106I

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

INTERVENTIONS:
Other: Phenotypic resistance measure — SDM experiments: Reverse transcriptase mutants of HIV-1 will be obtained by site-directed mutagenesis using specific primers introducing the expected mutations into plasmids pNL4.3 and CRF02_AG. HIV-1 stocks will be obtained by transfecting 293-T cells with the various HIV-1 molecular clones. 48 hours after transfection, the viral supernatants will be recovered, quantified for HIV-1p24gag antigen (Vidas BioMérieux) and frozen at -80°C.The single-cycle virus titers will be determined on HeLa-P4 cells in which the expression of b-galactosidase is inducible by the HIV Tat protein. Phenotypic analysis: creation of replication competent chimeric viruses through homologous recombination between patient or laboratory virus-derived PCR fragments and the corresponding NL4-3 vector where the whole Gag-PR, RT-RNaseH or IN coding regions have been deleted through inverse PCR. The susceptibility to Doravirine will be calculated through a single round infection assay in TZM-bl cells.

SUMMARY:
Objective. To study the impact of V106I mutation in the reverse transcriptase of HIV-1 on the activity of Doravirine.

Clinical hypotheses.

Doravirine shows a unique resistance pattern with a higher genetic barrier to resistance than other NNRTIs. In contrast to K103N or E138A, the prevalence of single mutations and/or combination of mutations against Doravirine is low. However, in a recent survey conducted in Spain the study investigators have found a V106Iprevalence similar to K103N and E138A. There is a clear need to understand the real impact of this mutation on Doravirine resistance.

DETAILED DESCRIPTION:
Testing for transmitted drug resistance (TDR) in the reverse transcriptase and protease in newly diagnosed patients with HIV is recommended by treatment guidelines. Currently clinical practice for first line treatment is moving to a test and treat approach. In this setting, Spanish GESIDA guidelines indicate that a first line protease (PI) or integrase (INI) inhibitor-based regimen may be started even if results from baseline resistance are yet not available. This indication is based on the very low prevalence of INI or PI TDR.

In Europe, TDR to NNRTIs has stabilized between 4-5%. Doravirine has a unique mutational pattern and its activity is affected by mutations that are usually not found at baseline as TDR (V106A/M, V108I, Y188L, G190S, F227 C/L/V, M230I/L, L234I, P236L Y318F and K103N/Y181C), as a recent European survey has already shown. In addition, these findings have been confirmed in a survey the study investigators have conducted in Spain. However, in this study the Stanford algorithm was used to evaluate clinical resistance to NNRTIs and, surprisingly found an unexpected high prevalence of resistance to Doravirine (as high as for first generation NNRTIs). Study investigators detected that resistance to Doravirine was mainly driven by V106I mutation, which Stanford scores as "low-level resistance".

MeditRes is a consortium of HIV clinical virologists from France (leader Anne-Genevieve Marcellin, Paris), Italy (leader Francesca Ceccerini-Silbesrtein, Rome, Spain (leader Federico García, Granada), Greece (leader Dimitrios Paraskevis, Athens) and Portugal (leader Perpetua Gomes, Lisbon). Each of these team leaders has access/coordinate local or national cohorts in their countries.

This study aims to investigate the prevalence of V106I TDR in patients joining the MEDITRES consortium during years 2018 and 2019. In patients carrying V106I in the background of a wild-type virus phenotypic resistance to Doravirine will be evaluated the Fold-Change (FC) will be calculated. In addition, Site Directed Mutagenesis (SDM) will be used to evaluate FC to Doravirine in the background of B and CRF02-AG subtypes. Patient recruitment will follow general recruitment procedures to be incorporated into each running cohorts currently contributing to MEDITRES (multicentre, prospective cohort of HIV-positive, antiretroviral-naïve subjects over 18 years of age, including both seroprevalent and seroconverter patients).

ELIGIBILITY:
Inclusion Criteria:

Antiretroviral-naïve subjects over 13 years of age, including both seroprevalent and seroconverter patients

Exclusion Criteria:

Patients with prior antiretroviral exposure

-

Ages: 13 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: HIV positive patients, newly diagnosed and naive to antiretroviral treatment
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-09-01 (Estimated); Primary Completion 2021-10-01 (Estimated); Study Completion 2022-05-01 (Estimated)

PRIMARY OUTCOMES:
Fold Change in resistance to Doravirine | Day 0
  Change in EC50 for resistance to Doravirine in the presence of V106I

REFERENCES:
- [Background] Panel de expertos de GeSIDA y Plan Nacional sobre el Sida. [GESIDA/National AIDS Plan: Consensus document on antiretroviral therapy in adults infected by the human immunodeficiency virus (Updated January 2015)]. Enferm Infecc Microbiol Clin. 2015 Oct;33(8):543.e1-43. doi: 10.1016/j.eimc.2015.03.016. Epub 2015 May 7. Spanish. PMID 25959461
- [Background] Hofstra LM, Sauvageot N, Albert J, Alexiev I, Garcia F, Struck D, Van de Vijver DAMC, Asjo B, Beshkov D, Coughlan S, Descamps D, Griskevicius A, Hamouda O, Horban A, Van Kasteren M, Kolupajeva T, Kostrikis LG, Liitsola K, Linka M, Mor O, Nielsen C, Otelea D, Paraskevis D, Paredes R, Poljak M, Puchhammer-Stockl E, Sonnerborg A, Stanekova D, Stanojevic M, Van Laethem K, Zazzi M, Zidovec Lepej S, Boucher CAB, Schmit JC, Wensing AMJ; SPREAD Program; Puchhammer-Stockl E, Sarcletti M, Schmied B, Geit M, Balluch G, Vandamme AM, Vercauteren J, Derdelinckx I, Sasse A, Bogaert M, Ceunen H, De Roo A, De Wit S, Echahidi F, Fransen K, Goffard JC, Goubau P, Goudeseune E, Yombi JC, Lacor P, Liesnard C, Moutschen M, Pierard D, Rens R, Schrooten Y, Vaira D, Vandekerckhove LPR, Van den Heuvel A, Van Der Gucht B, Van Ranst M, Van Wijngaerden E, Vandercam B, Vekemans M, Verhofstede C, Clumeck N, Van Laethem K, Beshkov D, Alexiev I, Lepej SZ, Begovac J, Kostrikis L, Demetriades I, Kousiappa I, Demetriou V, Hezka J, Linka M, Maly M, Machala L, Nielsen C, Jorgensen LB, Gerstoft J, Mathiesen L, Pedersen C, Nielsen H, Laursen A, Kvinesdal B, Liitsola K, Ristola M, Suni J, Sutinen J, Descamps D, Assoumou L, Castor G, Grude M, Flandre P, Storto A, Hamouda O, Kucherer C, Berg T, Braun P, Poggensee G, Daumer M, Eberle J, Heiken H, Kaiser R, Knechten H, Korn K, Muller H, Neifer S, Schmidt B, Walter H, Gunsenheimer-Bartmeyer B, Harrer T, Paraskevis D, Hatzakis A, Zavitsanou A, Vassilakis A, Lazanas M, Chini M, Lioni A, Sakka V, Kourkounti S, Paparizos V, Antoniadou A, Papadopoulos A, Poulakou G, Katsarolis I, Protopapas K, Chryssos G, Drimis S, Gargalianos P, Xylomenos G, Lourida G, Psichogiou M, Daikos GL, Sipsas NV, Kontos A, Gamaletsou MN, Koratzanis G, Sambatakou H, Mariolis H, Skoutelis A, Papastamopoulos V, Georgiou O, Panagopoulos P, Maltezos E, Coughlan S, De Gascun C, Byrne C, Duffy M, Bergin C, Reidy D, Farrell G, Lambert J, O'Connor E, Rochford A, Low J, Coakely P, O'Dea S, Hall W, Mor O, Levi I, Chemtob D, Grossman Z, Zazzi M, de Luca A, Balotta C, Riva C, Mussini C, Caramma I, Capetti A, Colombo MC, Rossi C, Prati F, Tramuto F, Vitale F, Ciccozzi M, Angarano G, Rezza G, Kolupajeva T, Vasins O, Griskevicius A, Lipnickiene V, Schmit JC, Struck D, Sauvageot N, Hemmer R, Arendt V, Michaux C, Staub T, Sequin-Devaux C, Wensing AMJ, Boucher CAB, van de Vijver DAMC, van Kessel A, van Bentum PHM, Brinkman K, Connell BJ, van der Ende ME, Hoepelman IM, van Kasteren M, Kuipers M, Langebeek N, Richter C, Santegoets RMWJ, Schrijnders-Gudde L, Schuurman R, van de Ven BJM, Asjo B, Kran AB, Ormaasen V, Aavitsland P, Horban A, Stanczak JJ, Stanczak GP, Firlag-Burkacka E, Wiercinska-Drapalo A, Jablonowska E, Maolepsza E, Leszczyszyn-Pynka M, Szata W, Camacho R, Palma C, Borges F, Paixao T, Duque V, Araujo F, Otelea D, Paraschiv S, Tudor AM, Cernat R, Chiriac C, Dumitrescu F, Prisecariu LJ, Stanojevic M, Jevtovic D, Salemovic D, Stanekova D, Habekova M, Chabadova Z, Drobkova T, Bukovinova P, Shunnar A, Truska P, Poljak M, Lunar M, Babic D, Tomazic J, Vidmar L, Vovko T, Karner P, Garcia F, Paredes R, Monge S, Moreno S, Del Amo J, Asensi V, Sirvent JL, de Mendoza C, Delgado R, Gutierrez F, Berenguer J, Garcia-Bujalance S, Stella N, de Los Santos I, Blanco JR, Dalmau D, Rivero M, Segura F, Elias MJP, Alvarez M, Chueca N, Rodriguez-Martin C, Vidal C, Palomares JC, Viciana I, Viciana P, Cordoba J, Aguilera A, Domingo P, Galindo MJ, Miralles C, Del Pozo MA, Ribera E, Iribarren JA, Ruiz L, de la Torre J, Vidal F, Clotet B, Albert J, Heidarian A, Aperia-Peipke K, Axelsson M, Mild M, Karlsson A, Sonnerborg A, Thalme A, Naver L, Bratt G, Karlsson A, Blaxhult A, Gisslen M, Svennerholm B, Bergbrant I, Bjorkman P, Sall C, Mellgren A, Lindholm A, Kuylenstierna N, Montelius R, Azimi F, Johansson B, Carlsson M, Johansson E, Ljungberg B, Ekvall H, Strand A, Makitalo S, Oberg S, Holmblad P, Hofer M, Holmberg H, Josefson P, Ryding U. Transmission of HIV Drug Resistance and the Predicted Effect on Current First-line Regimens in Europe. Clin Infect Dis. 2016 Mar 1;62(5):655-663. doi: 10.1093/cid/civ963. Epub 2015 Nov 29. PMID 26620652
- [Background] Soulie C, Santoro MM, Charpentier C, Storto A, Paraskevis D, Di Carlo D, Gennari W, Sterrantino G, Zazzi M, Perno CF, Calvez V, Descamps D, Ceccherini-Silberstein F, Marcelin AG. Rare occurrence of doravirine resistance-associated mutations in HIV-1-infected treatment-naive patients. J Antimicrob Chemother. 2019 Mar 1;74(3):614-617. doi: 10.1093/jac/dky464. PMID 30476106
- [Background] Guerrero-Beltran C, Martinez-Sanz J, Alvarez M, Olalla J, Garcia-Alvarez M, Iribarren JA, Masia M, Montero M, Garcia-Bujalance S, Blanco JR, Rivero M, Garcia-Fraile LJ, Espinosa N, Rodriguez C, Aguilera A, Vidal-Ampurdanes MC, Martinez M, Iborra A, Imaz A, Gomez-Sirvent JL, Peraire J, Portilla J, Caballero E, Alejos B, Garcia F, Moreno S; CoRIS. The algorithm used for the interpretation of doravirine transmitted drug resistance strongly influences clinical practice and guideline recommendations. J Antimicrob Chemother. 2020 May 1;75(5):1294-1300. doi: 10.1093/jac/dkaa009. PMID 32030406
- [Derived] Giammarino F, de Salazar A, Malet I, Vinuela L, Fuentes A, Saladini F, Bartolini N, Charpentier C, Lambert-Niclot S, Sterrantino G, Colao MG, Micheli V, Bertoli A, Fabeni L, Teyssou E, Delgado R, Falces-Romero I, Aguilera A, Gomes P, Paraskevis D, Santoro MM, Ceccherini-Silberstein F, Marcelin AG, Moreno C, Zazzi M, Garcia F. Prevalence and Phenotypic Susceptibility to Doravirine of the HIV-1 Reverse Transcriptase V106I Polymorphism in B and Non-B Subtypes. J Infect Dis. 2024 Jun 14;229(6):1796-1802. doi: 10.1093/infdis/jiae010. PMID 38206187